CLINICAL TRIAL: NCT02098850
Title: A Prospective International Study of Staphylococcus Aureus Bacteraemia in Adults by the International Staphylococcus Aureus Collaboration
Brief Title: Staphylococcus Aureus Bacteraemia in Adults
Acronym: ISAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Achim Kaasch, Dr. Achim Kaasch, University of Cologne
Other Study IDs: ISAC-01
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Staphylococcus aureus; bloodstream infection; bacteremia
MeSH Terms: conditions — Staphylococcal Infections; Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this evaluation is to record the management and outcome of adults with S.aureus bacteraemia (SAB) across multiple European, Asian and North American sites and to identify key quality indicators associated with improved outcome.

DETAILED DESCRIPTION:
Staphylococcus aureus (S. aureus) is one of the most common causes of bloodstream infections. Associated mortality has been reported to vary widely (4%-40%) although no obvious explanation for such variation has been identified.

Despite the existence of clinical guidelines, there is considerable variation in the management of S.aureus bacteraemia (SAB) between centres. Part of the variation in clinical management is due to the limited evidence base defining optimal therapy. Fewer than 1500 patients have been recruited to randomised controlled trials in the past 40 years; practice is therefore based largely on experience and observational studies.

The purpose of this evaluation is to record the management and outcome of adults with SAB across multiple European, Asian and North American sites. We aim to establish a broader knowledge base, identify key quality indicators associated with improved outcomes, and to provide comparator data to ensure that patients enrolled in randomized controlled trials are representative of bacteraemic S. aureus patients as a whole. All participating centres are experienced in the management of S. aureus bacteraemia and in conducting evaluations of current management practice and outcomes from S. aureus bacteraemia. Data is checked for plausibility by a centralized data quality control group.

ELIGIBILITY:
Inclusion Criteria:

* S. aureus (methicillin sensitive or resistant) isolated from one or more blood cultures

Exclusion Criteria:

* Recurrent episodes of S. aureus bloodstream infection
* Polymicrobial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in tertiary care hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 Days

SECONDARY OUTCOMES:
Length of hospital stay | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Kaasch, MD, Study Chair — University of Cologne
Locations (24):
- Germany (3):
  - Uniklinik Koln, Cologne, North Rhine-Westphalia
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Univeritatklinikum Schleswig-Holstein, Lübeck
- Seoul National University Bundang Hospital, Seoul, South Korea
- Spain (7):
  - Hospital San Pau, Barcelona
  - University Hospital Clinic de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Son Espases, Palma. Mallorca
  - Salamanca Hospital, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- Far Eastern Memorial Hospital, New Taipei City, Taiwan
- United Kingdom (12):
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Brighton and Sussex University Hospitals, Brighton
  - Cambridge University Hospitals, Cambridge
  - Hull and East Yorkshire Hospitals, Hull
  - Royal Liverpool and Broadgreen Hospital, Liverpool
  - Royal Free Hospital, London
  - Guy's and St Thomas', London
  - Kings College Hospital, London
  - University College London Hospital, London
  - Oxford University Hospitals, Oxford
  - Plymouth Hospitals, Plymouth
  - Portsmouth Hospitals, Portsmouth

REFERENCES:
- [Background] Kaasch AJ, Barlow G, Edgeworth JD, Fowler VG Jr, Hellmich M, Hopkins S, Kern WV, Llewelyn MJ, Rieg S, Rodriguez-Bano J, Scarborough M, Seifert H, Soriano A, Tilley R, Torok ME, Weiss V, Wilson AP, Thwaites GE; ISAC, INSTINCT, SABG, UKCIRG, and Colleagues. Staphylococcus aureus bloodstream infection: a pooled analysis of five prospective, observational studies. J Infect. 2014 Mar;68(3):242-51. doi: 10.1016/j.jinf.2013.10.015. Epub 2013 Nov 16. PMID 24247070